CLINICAL TRIAL: NCT05551091
Title: Glycomacropeptide as a Protein Supplement to Curb Hunger
Brief Title: Glycomacropeptide and Women's Health
Acronym: GMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1261; A074600 (Other: UW Madison); AG&LSC/NUTRITIONAL SCI/NUTRIT (Other: UW Madison); Protocol Version 8/11/2022 (Other: UW Madison)
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Obesity
Keywords: obesity; glucose tolerance; satiety; hunger; microbiome; amino acids; C-reactive protein
MeSH Terms: conditions — Obesity | interventions — caseinomacropeptide

STUDY DESIGN:
Intervention Model Description: Participants underwent measures of study outcomes at 4 time points: day 1 and day 7 of consuming GMP supplements twice daily (low-dose, 25 g before breakfast and dinner) and day 1 and day 7 of consuming GMP supplements thrice daily (high-dose, 25 g before breakfast, lunch and dinner). For each of the two baseline visits (day 1), participants consumed 300 kcal liquid breakfast meal tolerance test containing soy protein isolate, and then began the low-dose GMP or high-dose GMP for 7 days. On day 7 of each GMP diet, participants returned for a second GMP-based 300 kcal liquid breakfast meal tolerance test. Between the 2 weeks of GMP consumption, participants had a minimum washout period of 5 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMP 25 mg BID (Experimental): Investigators will conduct a pilot cross-over study in which 13 obese participants undergo measures of study outcomes: satiety hormones, glucose, amino acid and cytokine levels and changes in the fecal microbiota at baseline and after 7 days of consuming the supplement. On day one participants will consume a liquid soy breakfast, undergo study measures and then initiate GMP supplements twice a day (BID) x 7 days, with repeat study measures on day 7 of consuming the GMP supplement.
  Interventions: Dietary Supplement: glycomacropeptide (GMP)
- GMP 25 mg TID (Experimental): After a washout period, the same 13 participants will undergo repeated measures of study outcomes (satiety hormones, glucose, amino acid and cytokine levels and changes in the fecal microbiota). On day one subjects will consume a liquid soy breakfast, undergo study measures and then initiate GMP supplements thrice a day (TID) x 7 days, with repeat study measures on day 7 of consuming the GMP supplement.
  Interventions: Dietary Supplement: glycomacropeptide (GMP)

INTERVENTIONS:
Dietary Supplement: glycomacropeptide (GMP) — For each of the two baseline visits, women will consume a 300 calorie liquid breakfast meal tolerance test (MTT), eat a standard test lunch ad libitum with recording of food intake, and will then begin the low-dose GMP (25 g BID with meals) or high-dose GMP (25 g TID with meals) for 7 days. On day 7 of each GMP diet, women will come to the Clinical Research Unit (CRU) for a second breakfast MTT followed by lunch. All subjects will stop GMP products for 5-7 days (washout).

SUMMARY:
This is a study about how a dietary supplement containing a whey protein affects hormones controlling hunger and satiety (leptin and ghrelin) in postmenopausal women with a body mass index between 28 and 35 kg/m2. Participants can expect to be in study for 4 weeks.

DETAILED DESCRIPTION:
The purpose of this research study is to understand how a dietary supplement containing glycomacropeptide (GMP) affects blood sugar levels and hormones that regulate hunger and satiety. This study is being conducted to find new ways to help women lose weight and reduce their chance of getting diabetes.

ELIGIBILITY:
Inclusion Criteria:

* no more than 10 years past menopause as defined by the date of last menses, less than 90 years old, BMI of 28 to 35 kg/m2.

Exclusion Criteria:

* BMI>35 kg/m2, diabetes, and/or an active medical problem or condition that would interfere with study outcomes (malignancy, inflammatory condition, gastric bypass surgery or participation in another study)

Max Age: 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Glucose homeostasis | glucose levels 0, 15, 30, 45, 60, 90, 120 and 150 minutes postprandial
  Difference in glucose area under the curve after a soy versus a GMP liquid breakfast

SECONDARY OUTCOMES:
Ghrelin, a hormone regulating hunger and satiety | ghrelin levels 0, 15, 30, 45, 60, 90, 120 and 150 minutes postprandial
  Difference in ghrelin area under the curve after a soy versus a GMP liquid breakfast

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Hansen, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individuals who wish to obtain de-identified study data may contact Professor Ney.
Supporting Information: CSR
Time Frame: within 3 months of requesting the data
Access Criteria: Data sharing will commence after Institutional Review Board (IRB) approval to share the data, from University of Wisconsin and the individual's institution

REFERENCES:
- [Derived] Hansen KE, Murali S, Chaves IZ, Suen G, Ney DM. Glycomacropeptide Impacts Amylin-Mediated Satiety, Postprandial Markers of Glucose Homeostasis, and the Fecal Microbiome in Obese Postmenopausal Women. J Nutr. 2023 Jul;153(7):1915-1929. doi: 10.1016/j.tjnut.2023.03.014. Epub 2023 Apr 26. PMID 37116657